CLINICAL TRIAL: NCT06584279
Title: Diagnostic Value of MRI-targeted Plus Index-lesion-ipsilaterally Systematic Biopsy for Biopsy-naive Men At Risk of Prostate Cancer: a Prospective, Multicenter, Paired, Non-inferiority Trial
Brief Title: Diagnostic Value of MRI-targeted Plus Index-lesion-ipsilaterally Systematic Biopsy for Biopsy-naive Men At Risk of Prostate Cancer
Status: Recruiting | Type: Observational
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Hongqian Guo, Chief physician, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Other Study IDs: IUNU-PC-123
Record Dates: First submitted 2024-08-31; First posted 2024-09-04 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- prostate biopsy
  Interventions: Diagnostic Test: Biopsy of the prostate and pathological diagnosis

INTERVENTIONS:
Diagnostic Test: Biopsy of the prostate and pathological diagnosis — Whether the index-lesion-contralateral systematic biopsy was performed

SUMMARY:
Targeted and systematic biopsy stands as the prevalent diagnostic approach for prostate cancer. Despite its widespread use, this method is characterized by a high volume of needle biopsies. A refined approach, termed targeted and index-lesion-ipsilateral systematic biopsy, as one of targeted and regional systematic biopsy methods, aim to reduce the number of biopsy cores while maintaining an adequate positive rate. However, the absence of robust evidence necessitates further investigation. This study employs a prospective, multicenter, paired, non-inferiority design to assess the diagnostic efficacy of targeted and index-lesion-ipsilateral systematic prostate biopsy in comparison with the conventional targeted and systematic biopsy for the detection of clinically significant prostate cancer (csPCa). Eligible participants were identified as those with target lesions on prostate MRI, who subsequently underwent targeted and systematic prostate biopsies. The index lesion was defined as the one with the highest Prostate Imaging Reporting and Data System (PI-RADS) score; in cases of multiple lesions with identical PI-RADS scores, the lesion with the greatest diameter was prioritized. Post-biopsy pathological data were collected and evaluated using the International Society of Urological Pathology (ISUP) grading system, which classifies patients with a grade of 2 or higher as having csPCa. The study's primary outcome was to calculate the confidence interval for the difference in csPCa detection rates between the two biopsy methods under a paired design. This interval was then compared against a pre-specified non-inferiority margin to determine whether the targeted and index-lesion-ipsilateral systematic biopsy method is non-inferior to the standard targeted and systematic biopsy in detecting csPCa.

ELIGIBILITY:
Inclusion Criteria:

* Prostate specific antigen (PSA) >4 ng/ml;
* Prostate Imaging-Reporting and Data System (PI-RADS) score of any lesions on prostate magnetic resonance imaging ≥4 or PI-RADS score of lesions on prostate magnetic resonance imaging = 3 and prostate specific antigen density ≥0.1ng/cm3;
* accept prostate biopsy;

Exclusion Criteria:

* Prostate specific antigen>20ng/ml；
* the location of index lesion on prostate MRI is on the midline of the prostate and symmetrical on both sides;
* any contraindication of prostate biopsy;
* Previous prostate biopsy；
* Previous history of androgen deprivation therapy (ADT), pelvic radiotherapy, and other treatments；
* Previous history of transurethral prostatectomy (TURP)；

Ages: 60 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: biopsy-naive men at risk of prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 563 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Confidence interval for the difference in csPCa detection rate between targeted + index-lesion-ipsilaterally systematic biopsy and targeted + systematic biopsy for biopsy-naive men at risk of prostate cancer | 0.5-1 years

SECONDARY OUTCOMES:
additional value of index-lesion-contralaterally systematic biopsy | 0.5-1 years
pathological upgrade after radical prostatectomy | 0.5-1 years

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, China

IPD SHARING:
Plan to Share IPD: No